CLINICAL TRIAL: NCT00779415
Title: Long Term Prognosis of MRI Diagnosed Partial Thickness Tears of the Rotator Cuff
Status: Completed | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, April Armstrong, Associate Professor, Milton S. Hershey Medical Center
Other Study IDs: IRB26682EP
Record Dates: First submitted 2008-10-22; First posted 2008-10-24 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2015-02

CONDITIONS: Rotator Cuff Tear
Keywords: Partial Thickness; Rotator Cuff
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Partial Rotator Cuff Tear: Patients who presented from 1/1/02 to 12/31/06 to Hershey Medical Center with complaint of shoulder pain and were treated by the Orthopaedic Department

SUMMARY:
Patients diagnosed with partial thickness tears of the rotator cuff are sometimes surgically repaired, while other cases are not. It is unknown how patients fare over time without electing surgical repair and how outcomes differ by type of injury.

DETAILED DESCRIPTION:
We plan to conduct a retrospective cohort study to assemble a research database of all patients with shoulder pain from 1/1/02-12/31/06 presenting at the Hershey Medical Center. Participants will be identified using billing codes in the medical records office, with inclusion/exclusion criteria as described above. Data extraction will include medical record number, demographic data (age, race/ethnicity, sex, insurance type), pre-fracture functional status, pre-admission residence, medical co-morbidities, prior hospitalization within 30 days, abnormal clinical findings on admission, shoulder score, pain score, range of motion score, type of diagnosis (partial tear, full thickness tear, tendonitis, shoulder pain), occupation, past medical history, physical therapy and duration of physical therapy, cigarette/cigar use, drug use, alcohol use, treatment protocols (anti-inflammatory medication, injections, etc.), and complaints by patient of pain status.

ELIGIBILITY:
Inclusion Criteria:

* Patients examined at the Hershey Medical Center from 1/1/02-12/31/06 with a documented MRI report of a partial thickness tear of the rotator cuff that was treated non-operatively.

Exclusion Criteria:

* Full thickness tear of the rotator cuff, surgically repaired rotator cuff, and patients who do not fit criteria listed in inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who presented from 1/1/02 to 12/31/06 to Hershey Medical Center with complaint of shoulder pain and were treated by the Orthopaedic Department.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2008-07; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Creation of a database of patients with partial rotator cuff tears documented by MRI. | Retrospective review from 1/1/02 to 12/31/06, four years.

CONTACTS AND LOCATIONS:
Overall Officials: April D Armstrong, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State College of Medicine, Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Background] Nakatani T, Fujita K, Iwasaki Y, Sakai H, Kurosaka M. MRI-negative rotator cuff tears. Magn Reson Imaging. 2003 Jan;21(1):41-5. doi: 10.1016/s0730-725x(02)00630-6. PMID 12620544
- [Background] Ogilvie-Harris DJ, Wiley AM. Arthroscopic surgery of the shoulder. A general appraisal. J Bone Joint Surg Br. 1986 Mar;68(2):201-7. doi: 10.1302/0301-620X.68B2.3958003.
- [Background] Yamanaka K, Matsumoto T. The joint side tear of the rotator cuff. A followup study by arthrography. Clin Orthop Relat Res. 1994 Jul;(304):68-73. PMID 8020236
- [Background] Yamaguchi K, Tetro AM, Blam O, Evanoff BA, Teefey SA, Middleton WD. Natural history of asymptomatic rotator cuff tears: a longitudinal analysis of asymptomatic tears detected sonographically. J Shoulder Elbow Surg. 2001 May-Jun;10(3):199-203. doi: 10.1067/mse.2001.113086. PMID 11408898
- [Background] Yamaguchi K, Ditsios K, Middleton WD, Hildebolt CF, Galatz LM, Teefey SA. The demographic and morphological features of rotator cuff disease. A comparison of asymptomatic and symptomatic shoulders. J Bone Joint Surg Am. 2006 Aug;88(8):1699-704. doi: 10.2106/JBJS.E.00835. PMID 16882890